## Daily Delivery and Supervision of Psychotropic Medications for High-Risk Patients with Severe and Persistent Mental Illness

**Document date:** January 17, 2018

## **Analyses**

A description of the statistical methods to be employed, including timing of any planned analysis(ses). Collected data would be analyzed for significant outcomes comparing before and after (a two year total time frame from pre-index date to post-index date) findings for:

- number of days/visits spent with crisis services (ED & CRC),
- hospital visits/admissions (length of stay) and
- number of incarcerations (as a dependent variable)

These data would be entered into a multivariate analysis of covariance (MANCOVA) model or similar multi-level model with baseline or study time, age and gender as the independent variables. Descriptive statistics would be used to elaborate on patient satisfaction and other variables of interest. Preliminary cost analysis will also be undertaken in anticipation of calculating a net benefit for the daily dispensing services.

The number of subjects planned to be studied. N = 32

The level of significance to be used for any differences p < 0.05

Criteria for the termination of the study. Timeframe of study = approximately one year.

Procedure for accounting for missing, unused, and spurious data. Cleaning data, missing data analyses and manual review of data collected etc.

Procedures for reporting any deviation(s) from the original statistical plan (any deviation(s) from the original statistical plan should be described and justified in protocol and/or in the final report, as appropriate).

All deviations from the statistical plan will be based on the quality of data collected during the study and will be filed as amendments to the protocol with the Ethics Board.

The selection of subjects to be included in the analyses (e.g., evaluable subjects). Participants who are currently part of the Forensics program and who are enrolled in the daily dispensing program and have participated in the program for at least one month will be included in the analyses